CLINICAL TRIAL: NCT06095141
Title: Cisplatin Based Regimen to Patients With Advanced Pancreatic Cancer and Homologous Recombination Deficiency
Brief Title: Cisplatin to Patients With Pancreatic Cancer and Homologous Recombination Deficiency
Acronym: PTCA199-6
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-6
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Adenocarcinoma; Homologous Recombination Deficiency
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin (Experimental): Cisplatin 25 mg/m2, ivgtt, 30 min, D1, 8.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 25 mg/m2, ivgtt, 30 min, D1, 8. The administration of other chemotherapeutic agents including gemcitabine, nab-paclitaxel, fluorouracil, irinotecan, capecitabine is applied according to the National Comprehensive Cancer Network (NCCN) guideline. PARP inhibitor will be recommended to patients with platinum-sensitive metastatic PDAC after six months of cisplatin based regimen.

SUMMARY:
The purpose of this study is to evaluate the efficacy of cisplatin based regimen to patients with advanced pancreatic cancer and homologous recombination deficiency.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. In 2011, the PRODIGE trial has shown that oxaliplatin, irinotecan, fluorouracil, and leucovorin (FOLFIRINOX) was associated with a survival advantage but had increased toxicity.

Defects in DNA damage response (DDR) genes causing homologous recombination deficiency (HRD) identify a clinically relevant subgroup of patients with PDAC, with both therapeutic and preventative implications. Accumulating evidence from nonrandomized and randomized clinical trials suggests HRD as a putative biomarker of therapeutic response for platinum-based chemotherapy in patients with advanced PDAC. Within HRD, germline variants in BRCA1 and BRCA2 are associated with improved progression-free survival in patients with platinum-sensitive metastatic PDAC treated with the poly (ADP-ribose) polymerase (PARP) inhibitor (PARPi) olaparib as maintenance therapy. Interestingly, based on preclinical evidence and phase II nonrandomized clinical trials, additional non-BRCA HRD aberrations may predict sensitivity to PARPi with other therapeutic strategies targeting DDR currently under clinical investigation (including immunotherapy, ATM, ATR, and PALB2 inhibitors). However, the efficacy of cisplatin based regimen as a second line treatment for patients with HRD has not been systematically studied.

The purpose of this study is to evaluate the efficacy of cisplatin based regimen on improving the progression-free survival (PFS) of advanced pancreatic cancer patients who harbor germline or somatic homologous recombination deficiency. These patients are resistant to at least one line of systemic chemotherapy. PFS, objective response rate (ORR), overall survival (OS) and disease control rate (DCR) are measured every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed advanced pancreas adenocarcinoma.
* Tumor progression after at least one line of chemotherapy.
* Genetic or molecular test confirmed the presence of homologous recombination deficiency.
* Presence of at least of one measurable lesion in agreement to RECIST criteria.
* The expected survival ≥ 3 months.
* Adequate organ performance based on laboratory blood tests.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Pregnant or nursing women.
* Primary pancreatic cancer.
* Patients who have received platinum or PARPi treatment.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
* Renal insufficiency or dialysis
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
* Patients who are allergic to cisplatin or other platinum drugs.
* Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival, PFS | At the end of Cycle 1 (each cycle is 21 days)
  PFS of subjects from recruiting to the time of disease progression

SECONDARY OUTCOMES:
objective response rate (ORR) | At the end of Cycle 1 (each cycle is 21 days)
  CR + PR
disease control rate (DCR) | At the end of Cycle 1 (each cycle is 21 days)
  CR + PR + SD
Overall survival，OS | At the end of Cycle 1 (each cycle is 21 days)
  OS of subjects from recruiting to the time of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Reilly EM, Lee JW, Zalupski M, Capanu M, Park J, Golan T, Tahover E, Lowery MA, Chou JF, Sahai V, Brenner R, Kindler HL, Yu KH, Zervoudakis A, Vemuri S, Stadler ZK, Do RKG, Dhani N, Chen AP, Kelsen DP. Randomized, Multicenter, Phase II Trial of Gemcitabine and Cisplatin With or Without Veliparib in Patients With Pancreas Adenocarcinoma and a Germline BRCA/PALB2 Mutation. J Clin Oncol. 2020 May 1;38(13):1378-1388. doi: 10.1200/JCO.19.02931. Epub 2020 Jan 24. PMID 31976786
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963